CLINICAL TRIAL: NCT02914210
Title: Virtual Exercise Rehabilitation In-home Therapy: A Randomized Study (VERITAS)
Brief Title: Virtual vs. Traditional Physical Therapy Following Total Knee Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Reflexion Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00074409
Record Dates: First submitted 2016-09-15; First posted 2016-09-26 (Estimated); Results first posted 2020-01-18 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Total Knee Replacement
Keywords: TKR; TKA; Knee; Surgery; Replacement; Rehabilitation; Virtual; Physical Therapy; Telerehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual physical therapy (Other): Virtual physical therapy rehabilitation program (VERA) used in the home with care planning and remote support and monitoring by physical therapists
  Interventions: Device: Virtual physical therapy rehabilitation program
- Traditional physical therapy (Other): No intervention. Standard home health physical therapy and/or outpatient clinic physical therapy as prescribed.
  Interventions: Other: No intervention

INTERVENTIONS:
Device: Virtual physical therapy rehabilitation program — Virtual Exercise Rehabilitation Assistant (VERA), a virtual physical therapy delivery system installed in patient's home
  Arms: Virtual physical therapy
Other: No intervention — Traditional physical therapy delivered in clinic or via home-health visits
  Arms: Traditional physical therapy

SUMMARY:
The goals of this research study are the following:

1. To compare the effects of tele-rehabilitation-supported physical therapy versus traditional home and/or clinic-based physical therapy for total knee replacement (TKR) on 90-day health service use costs.
2. To compare tele-rehabilitation-supported physical therapy and traditional physical therapy on patient-centered outcomes
3. To explore whether individual patient characteristics are associated with differential improvement from 6 to 12 weeks assessed by patient-reported outcomes.

DETAILED DESCRIPTION:
This study will compare the effects on health service use costs of tele-rehabilitation-supported physical therapy versus traditional home and/or clinic-based physical therapy following total knee replacement (TKR) surgery. It will also examine standard post-surgical clinical measures to confirm non-inferiority of outcomes between groups. A total of 300 patients will receive standard pre- and post-surgical medical care from their healthcare providers, and be randomized to receive pre-surgery rehabilitation exercises ("pre-hab") and post-discharge physical therapy provided via either a home-based tele-rehabilitation platform (intervention group, n=150) or home-health and clinic-based physical therapy regimen (control group, n=150). Data will be collected by sites at enrollment, baseline, hospital discharge, and 6 weeks following surgery. Patients will complete telephone surveys regarding their health and knee function at baseline, 6 weeks, and 3 months after surgery. Patients will also keep a diary from hospital discharge through 3 months documenting healthcare utilization and progress toward a personal recovery goal. Diary information will be collected over the phone concurrently with administration of the 6-week and 3-month surveys. The episode for analysis will be from surgery through 3 months post-discharge, in alignment with the Centers for Medicare and Medicaid Services Comprehensive Care for Joint Replacement (CJR) bundled payment model. Physical risks or benefits to patients for participating in this study are as expected from standard pre- and post-surgical physical therapy associated with total knee replacement surgery. The low risk of loss of confidentiality for all subjects will be minimized using appropriate safeguards.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age
2. Scheduled to have a non-traumatic TKR
3. Can be enrolled a minimum of 10 days prior to surgery (in-person visit)
4. Have a Risk Assessment and Prediction Tool (RAPT) score of ≥ 6 indicating expected discharge home after surgical hospitalization

Exclusion Criteria:

1. Unable or unwilling to provide informed consent, including but not limited to cognitive or language barriers (comprehension)
2. Scheduled for staged bilateral TKR
3. Living in a nursing home prior to surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janet Bettger, ScD, Principal Investigator — Duke Clinical Research Institute, Duke Dept of Orthopaedic Surgery
Locations (4):
- United States (4):
  - University of North Carolina Orhthopedics, Chapel Hill, North Carolina
  - Duke Orthopaedics, Durham, North Carolina
  - Greensboro Orthopedics, Greensboro, North Carolina
  - Raleigh Orthopaedics, Raleigh, North Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Virtual Physical Therapy | Traditional Physical Therapy
Started | 153 | 153
Completed | 143 | 144
Not Completed | 10 | 9

BASELINE CHARACTERISTICS:
Population: Enrolled patients excluding those found to be ineligible after enrollment and prior to surgery
Groups:
- Total: Total of all reporting groups
Arm/Group | Virtual Physical Therapy | Traditional Physical Therapy | Total
Number analyzed (Participants) | 151 | 153 | 304
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.4 (7.7) | 65.1 (9.2) | 65.2 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90 | 100 | 190
  Male | 61 | 53 | 114
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 128 | 119 | 247
  Race: Black | 16 | 28 | 44
  Race: Other | 2 | 3 | 5
  Race: Multiple | 4 | 3 | 7
  Race: Missing | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino Ethnicity: Yes | 4 | 0 | 4
  Hispanic or Latino Ethnicity: No or Not Reported | 147 | 153 | 300
Region of Enrollment [Number; unit: participants]
  United States | 151 | 153 | 304
RAPT Score [Mean (Standard Deviation); unit: units on a scale] — Standardized Risk Assessment and Prediction Tool (RAPT) used to predict likely discharge destination in patients undergoing elective hip or knee replacement. Scores range from 1-12. Score < 6 indicates likely discharge to inpatient rehab; these patients were not eligible for enrollment. Score of 6 or higher indicates likely discharge to home, with or without supportive services such as home health.
  units on a scale | 10.1 (1.3) | 9.7 (1.6) | 9.9 (1.4)

OUTCOME MEASURES:

1. Primary Outcome: Cost Difference in US Dollars
Description: Difference in total health service use costs at 12-weeks postoperative between patients who receive tele-rehab-supported PT versus traditional home and/or clinic-based PT for TKR.
Time Frame: 12 weeks
Population: Patients randomized and receiving eligible surgery, and completing the study through 12 weeks post surgery.
Measure: Median (Inter-Quartile Range); unit: US Dollars
Arm/Group | Virtual Physical Therapy | Traditional Physical Therapy
Number analyzed (Participants) | 143 | 144
US Dollars | 1050.00 [900.00 to 1200.00] | 2805.00 [1644.50 to 4505.00]

2. Secondary Outcome: Knee Injury and Osteoarthritis Outcome Score (KOOS)
Description: Survey regarding health [Knee Injury and Osteoarthritis Outcome Score (KOOS)] for pain, symptoms, activities of daily living, function in sports and recreation, and knee-related quality of life (QOL) at 6 weeks and 12 weeks, scored from 0 to 100. Higher score indicates better outcomes.
Time Frame: 6 weeks and 12 weeks
Population: Patients randomized and receiving eligible surgery, completing study through 12 weeks, and providing complete responses to survey questions
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Virtual Physical Therapy | Traditional Physical Therapy
Number analyzed (Participants) | 143 | 144
score on a scale
  6 weeks | 61.0 (11.5) | 61.8 (13.5)
  12 weeks | 69.6 (12.1) | 67.2 (14.3)

3. Secondary Outcome: Range of Motion
Description: Knee range of motion [lower (extension) and upper range of motion (flexion)] at 6 weeks
Time Frame: 6 weeks
Population: Patients randomized and receiving eligible surgery, completing study through 12 weeks, and having range of motion measured at specified time point.
Measure: Mean (Standard Deviation); unit: degrees from parallel to floor
Arm/Group | Virtual Physical Therapy | Traditional Physical Therapy
Number analyzed (Participants) | 143 | 144
degrees from parallel to floor
  Knee Extension (straight leg) | 2.5 (3.6) | 2.9 (3.4)
  Knee Flexion (bent leg) | 114.5 (15.3) | 111.4 (16.0)

4. Secondary Outcome: 10-meter Gait Speed
Description: Gait speed 6 weeks after surgery
Time Frame: 6 weeks
Population: Patients randomized and receiving eligible surgery, completing study through 12 weeks, and having gait speed measured.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Virtual Physical Therapy | Traditional Physical Therapy
Number analyzed (Participants) | 143 | 144
minutes | 1.0 (0.3) | 1.0 (0.3)

5. Secondary Outcome: Pain Score
Description: Non-inferiority safety endpoint: pain score at 12 weeks. Measured on scale from 0 to 10, with 0 being no pain and 10 being worst pain imaginable.
Time Frame: 12 weeks
Population: Patients randomized and receiving eligible surgery, completing study through 12 weeks, and responding to survey question regarding pain.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Virtual Physical Therapy | Traditional Physical Therapy
Number analyzed (Participants) | 143 | 144
score on a scale | 2.7 (2.0) | 3.0 (2.6)

6. Secondary Outcome: Report of Falls
Description: Any fall reported between hospital discharge and 12-week follow-up (yes/no)
Time Frame: 12 weeks
Population: Patients randomized and receiving eligible surgery, completing study through 12 weeks, and answering survey question regarding falls.
Measure: Number; unit: percentage of patients
Arm/Group | Virtual Physical Therapy | Traditional Physical Therapy
Number analyzed (Participants) | 143 | 144
percentage of patients | 19.4 | 14.6

7. Secondary Outcome: Re-hospitalization
Description: Re-hospitalizations since hospital discharge (total count)
Time Frame: 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: number of rehospitalizations per patient
Arm/Group | Virtual Physical Therapy | Traditional Physical Therapy
Number analyzed (Participants) | 143 | 144
number of rehospitalizations per patient | 0.1 (0.3) | 0.2 (0.5)

8. Other Pre Specified Outcome: Knee Injury and Osteoarthritis Outcome Score (KOOS) Sub-domain Scores
Description: Scores in KOOS sub-domains of pain, symptoms, activities of daily living (ADL), sports and recreation, and quality of life (QOL). Each sub-domain score can be normalized to values ranging from 0 to 100. Higher scores denote better outcomes.
Time Frame: 6 weeks and 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Virtual Physical Therapy | Traditional Physical Therapy
Number analyzed (Participants) | 143 | 144
score on a scale
  Pain (6 weeks) | 66.6 (15.6) | 68.7 (17.1)
  Symptoms (6 weeks) | 54.7 (11.5) | 53.9 (11.8)
  Function/Daily Living (6 weeks) | 76.4 (13.9) | 75.7 (16.6)
  Sports/Recreation (6 weeks) | 51.2 (29.4) | 50.2 (31.0)
  Quality of Life (6 weeks) | 46.5 (18.7) | 50.5 (19.6)
  Pain (12 weeks) | 78.4 (14.0) | 76.7 (17.5)
  Symptoms (12 weeks) | 54.9 (12.2) | 53.9 (11.1)
  Function/Daily Living (12 weeks) | 82.7 (13.6) | 80.9 (17.7)
  Sports/Recreation (12 weeks) | 75.6 (109.2) | 61.5 (28.3)
  Quality of Life (12 weeks) | 61.8 (18.8) | 58.3 (20.0)

9. Other Pre Specified Outcome: Physical Activity
Description: Physical activity (duration of moderate exercise in total minutes per week)
Time Frame: 6 weeks and 12 weeks
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: minutes per week
Arm/Group | Virtual Physical Therapy | Traditional Physical Therapy
Number analyzed (Participants) | 143 | 144
minutes per week
  6 weeks | 40 [0 to 150] | 4 [0 to 90]
  12 weeks | 60 [0 to 150] | 60 [0 to 120]

10. Other Pre Specified Outcome: Return to Work
Description: Return to work (yes, modified schedule, or no) for those who stopped working prior to surgery
Time Frame: 6 weeks and 12 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Virtual Physical Therapy | Traditional Physical Therapy
Number analyzed (Participants) | 68 | 65
Participants
  6 weeks: Yes | 15 | 14
  6 weeks: Modified Schedule | 17 | 18
  6 weeks: No | 36 | 32
  6 weeks: Not recorded | 0 | 1
  12 weeks: Yes | 41 | 42
  12 weeks: Modified Schedule | 9 | 12
  12 weeks: No | 13 | 11
  12 weeks: Not recorded | 5 | 0

11. Other Pre Specified Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS) - Mental Health (MH) Score
Description: PROMIS mental health score at 12 weeks, on a scale of 0 to 20 with higher scores indicating better mental health.
Time Frame: 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Virtual Physical Therapy | Traditional Physical Therapy
Number analyzed (Participants) | 143 | 144
score on a scale | 16.6 (2.5) | 16.1 (3.2)

12. Other Pre Specified Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS) - Physical Health (PH) Score
Description: PROMIS physical health score at 12 weeks, on a scale of 0 to 20, with higher scores indicating better physical health.
Time Frame: 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Virtual Physical Therapy | Traditional Physical Therapy
Number analyzed (Participants) | 143 | 144
score on a scale | 15.3 (2.4) | 14.8 (2.8)

13. Other Pre Specified Outcome: Satisfaction With Physical Function
Description: Score on Satisfaction with Physical Function questionnaire through 12 weeks after surgery, on a scale of 0 to 6, with 6 being higher satisfaction.
Time Frame: 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Virtual Physical Therapy | Traditional Physical Therapy
Number analyzed (Participants) | 143 | 144
score on a scale | 4.9 (1.3) | 4.9 (1.2)

14. Other Pre Specified Outcome: Satisfaction With Tele-rehab Platform
Description: Satisfaction with tele-rehab platform, on scale of 0 to 10, with 10 being highly satisfied.
Time Frame: 12 weeks
Population: Patients randomized and receiving eligible surgery, completing study through 12 weeks, using the virtual platform at least once, and providing response to survey question.
Measure: Number; unit: percentage of participants
Arm/Group | Virtual Physical Therapy
Number analyzed (Participants) | 143
percentage of participants
  Promoters (score 9-10) | 83.3
  Detractors (score 0-6) | 9.5
  Neutral (score 7-8) | 7.2

ADVERSE EVENTS:
Time Frame: Mortality at discharge from surgical hospitalization.
Description: Mortality was assessed at hospital discharge only, using available medical records. No other adverse events were assessed since this was a study of cost savings between marketed virtual physical therapy assistant and traditional clinic/home-health-based physical therapy.
Arm/Group | Virtual Physical Therapy | Traditional Physical Therapy
All-Cause Mortality (participants affected / at risk) | 0/143 | 0/144
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2017-03-02): https://cdn.clinicaltrials.gov/large-docs/10/NCT02914210/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-08): https://cdn.clinicaltrials.gov/large-docs/10/NCT02914210/SAP_001.pdf
  • Informed Consent Form (2016-08-17): https://cdn.clinicaltrials.gov/large-docs/10/NCT02914210/ICF_002.pdf